CLINICAL TRIAL: NCT01299376
Title: A Phase III, Randomized, Active-Comparator Controlled Clinical Trial to Study the Efficacy and Safety of MK-0954E in Japanese Patients With Essential Hypertension Uncontrolled With MK-954H (L50/H12.5 mg) [PREMINENT®] and an Open-label, Long-term Clinical Trial to Study the Safety of MK-0954E
Brief Title: MK-0954E Phase III Long-Term Study in Participants With Hypertension (MK-0954E-356)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0954E-356
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Results first posted 2017-01-26 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-07

CONDITIONS: Hypertension
Keywords: Essential hypertension; Antihypertensive agents; Blood pressure; Uncontrolled hypertension
MeSH Terms: conditions — Hypertension; Essential Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- L50/H12.5/A5→L50/H12.5/A5 (Experimental): One combination tablet containing L50 mg, H12.5 mg, and A5 mg, orally, once daily, for up to 8 weeks (double-blind treatment period). Participants continue with once daily L50/H12.5/A5 for 44 weeks during open label extension.
  Interventions: Drug: L50/H12.5/A5; Drug: Placebo to L50/H12.5
- L50/H12.5→L50/H12.5/A5 (Active Comparator): One combination tablet containing L50 mg and H12.5 mg, orally, once daily, for up to 8 weeks during double-blind treatment period. Participants then receive once daily L50/H12.5/A5 for 44 weeks during open-label extension
  Interventions: Drug: L50/H12.5; Drug: Placebo to L50/H12.5/A5

INTERVENTIONS:
Drug: L50/H12.5/A5
  Other Names: MK-0954E
  Arms: L50/H12.5/A5→L50/H12.5/A5
Drug: L50/H12.5
  Other Names: MK-0954H
  Arms: L50/H12.5→L50/H12.5/A5
Drug: Placebo to L50/H12.5/A5
  Arms: L50/H12.5→L50/H12.5/A5
Drug: Placebo to L50/H12.5
  Arms: L50/H12.5/A5→L50/H12.5/A5

SUMMARY:
This study has two parts. In the first part, the efficacy and safety MK-0954E (losartan potassium 50 mg [L50] (+) hydrochlorothiazide 12.5 mg [H12.5] (+) amlodipine besylate 5mg [A5]) will be evaluated and compared to the efficacy and safety of MK-0954H (L50/H12.5) in Japanese participants. In the second part, the safety and tolerability of long-term use of open-label MK-0954E in participants with hypertension will be evaluated. The primary hypothesis is that MK-0954E is more effective in lowering mean trough sitting diastolic blood pressure (SiDBP) after 8 weeks of treatment compared to MK-954H (L50/H12.5 mg) in Japanese participants with essential hypertension who are not adequately controlled following a 8-week treatment with filter period study drug of MK-954H.

ELIGIBILITY:
Inclusion criteria:

* Participant has a diagnosis of essential hypertension
* Participant is being treated with a single, or dual combination treatment for hypertension and will be able to discontinue the prior antihypertensive medication
* Participant has a mean trough SiDBP of ≥ 90 mmHg and < 110 mmHg
* Participant has a mean trough SiSBP of ≥ 140 mmHg and < 200 mmHg
* Participant has no clinically significant abnormality at screening visit

Exclusion criteria:

* Participant is currently taking >2 antihypertensive medications
* Participant has a history of significant multiple and/or severe allergies to ingredients of Nu-Lotan or Preminent, amlodipine or dihydropyridine drug and thiazide drug or related drug (i.e., sulfonamide-containing "chlortalidone" medicines)
* Participant is, at the time of signing informed consent, a user of recreational or illicit drugs or has had a recent history within the last year of drug or alcohol abuse or dependence
* Participant is pregnant or breastfeeding, or expecting to conceive OR the pregnancy test is positive at screening visit (Visit 1)
* Participant is currently participating or has participated in a study with an investigational compound or device within 30 days of signing informed consent

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2011-01-24 (Actual); Primary Completion 2011-11-16 (Actual); Study Completion 2012-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Rakugi H, Tsuchihashi T, Shimada K, Numaguchi H, Nishida C, Yamaguchi H, Shirakawa M, Azuma K, Fujita KP. Efficacy and safety of fixed-dose losartan/hydrochlorothiazide/amlodipine combination versus losartan/hydrochlorothiazide combination in Japanese patients with essential hypertension. Clin Exp Hypertens. 2015;37(3):260-6. doi: 10.3109/10641963.2014.954712. Epub 2014 Oct 1. PMID 25271811

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants received single-blind losartan 50 mg (L50)/hydrochlorothiazide 12.5 mg (H12.5) and placebo for L50/H12.5/amlodipine 5 mg (A5) during 8-week Filter Period. A total of 510 entered the Filter Period and 286 were randomly assigned to 1 of the 2 treatment arms for the Double-blind Treatment Period.
Groups:
- L50/H12.5/A5→L50/H12.5/A5: One combination tablet containing L50 mg, H12.5 mg, and A5 mg, orally, once daily, for up to 8 weeks (double-blind treatment period). Participants continue with once daily L50/H12.5/A5 for 44 weeks during open-label extension.
Period: Double-blind Treatment (Weeks 1 to 8)
Arm/Group | L50/H12.5/A5→L50/H12.5/A5 | L50/H12.5→L50/H12.5/A5
Started | 141 | 145
Completed | 134 | 133
Not Completed | 7 | 12
Not completed — Adverse Event | 1 | 2
Not completed — Lack of Efficacy | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Blood Pressure/Potassium Criteria Met | 4 | 7
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Period: Extension (Weeks 9 to 52)
Arm/Group | L50/H12.5/A5→L50/H12.5/A5 | L50/H12.5→L50/H12.5/A5
Started | 134 | 133
Completed | 124 | 118
Not Completed | 10 | 15
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Adverse Event | 2 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Blood Pressure/Potassium Criteria Met | 4 | 9
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | L50/H12.5/A5→L50/H12.5/A5 | L50/H12.5→L50/H12.5/A5 | Total
Number analyzed (Participants) | 141 | 145 | 286
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.9 (9.1) | 56.3 (9.7) | 55.1 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 34 | 67
  Male | 108 | 111 | 219

OUTCOME MEASURES:

1. Primary Outcome: Change in Trough Sitting Diastolic Blood Pressure (SiDBP)-Double-Blind Treatment Period
Description: Sitting diastolic blood pressure was measured by automated sphygmomanometer pre-dose on Day 1 (baseline) and at 24 ± 2 hours after the last study drug administration at Week 8. The difference between the baseline and Week 8 assessments was calculated and summarized by treatment arm.
Time Frame: Baseline and Week 8
Population: All participants that received at least one dose of study treatment during double-blind treatment period , had at least 1 post-randomization observation for the analysis endpoint, and had baseline data
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Groups:
- L50/H12.5/A5: One combination tablet containing L50 mg H12.5 mg and A5, orally, once daily, for up to 8 weeks during double-blind treatment period.
- L50/H12.5: One combination tablet containing L50 mg and H12.5 mg, orally, once daily, for up to 8 weeks during double-blind treatment period.
Arm/Group | L50/H12.5/A5 | L50/H12.5
Number analyzed (Participants) | 141 | 144
mmHg | -12.1 [-13.3 to -10.9] | -6.2 [-7.4 to -5.0]
Statistical Analysis 1: Comparison: L50/H12.5/A5 vs L50/H12.5; Test type: Superiority or Other; p < 0.001, Contrained Longitudinal Data Analysis; Model including treatment, time and the interaction of time by treatment with a restriction of the same baseline mean across treatment groups; Difference in Least-squares Means = -5.9, 95% CI 2-sided [-7.5 to -4.2]

2. Primary Outcome: Percentage of Participants Who Experience 1 or More Adverse Events (AEs)- Double-Blind Treatment Period
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. The percentage of participants who experienced at least 1 AE during the 8-week double-blind treatment period were summarized by study drug received.
Time Frame: up to Week 8
Population: All randomized participants who received at least 1 dose of study drug during double-blind treatment period.
Measure: Number; unit: Percentage of Participants
Arm/Group | L50/H12.5/A5 | L50/H12.5
Number analyzed (Participants) | 141 | 145
Percentage of Participants | 27.0 | 29.7

3. Primary Outcome: Percentage of Participants Who Experience 1 or More Drug-Related AEs- Double-Blind Treatment Period
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. Percentage of participants that experienced at least 1 AE that was reported as possibly, probably, or definitely related to the study drug by the investigator during the 8-week double-blind treatment period were summarized by study drug received.
Time Frame: up to Week 8
Population: All randomized participants who received at least 1 dose of study drug during double-blind treatment period.
Measure: Number; unit: Percentage of Participants
Arm/Group | L50/H12.5/A5 | L50/H12.5
Number analyzed (Participants) | 141 | 145
Percentage of Participants | 12.1 | 14.5

4. Primary Outcome: Percentage of Participants Who Experience 1 or Serious Adverse Events (SAEs)- Double-Blind Treatment Period
Description: An SAE is any AE occurring at any dose or during any use of Sponsor's product that does the following: results in death; is life threatening; results in persistent or significant disability/incapacity; results in or prolongs an existing inpatient hospitalization; is a congenital anomaly/birth defect; is a cancer; is associated with an overdose; is another important medical event. The percentage of participants who experienced at least 1 SAE during the 8-week double-blind treatment period were summarized by study drug received.
Time Frame: up to Week 8
Population: All randomized participants who received at least 1 dose of study drug during double-blind treatment period.
Measure: Number; unit: Percentage of Participants
Arm/Group | L50/H12.5/A5 | L50/H12.5
Number analyzed (Participants) | 141 | 145
Percentage of Participants | 0.7 | 1.4

5. Primary Outcome: Percentage of Participants Who Experience 1 or More Drug-Related Serious Adverse Events (SAEs)- Double-Blind Treatment Period
Description: An SAE is any AE occurring at any dose or during any use of Sponsor's product that does the following: results in death; is life threatening; results in persistent or significant disability/incapacity; results in or prolongs an existing inpatient hospitalization; is a congenital anomaly/birth defect; is a cancer; is associated with an overdose; is another important medical event. Percentage of participants that experienced at least 1 SAE that was reported as possibly, probably, or definitely related to the study drug by the investigator during the 8-week double-blind treatment period were summarized by study drug received.
Time Frame: up to Week 8
Population: All randomized participants who received at least 1 dose of study drug during double-blind treatment period.
Measure: Number; unit: Percentage of Participants
Arm/Group | L50/H12.5/A5 | L50/H12.5
Number analyzed (Participants) | 141 | 145
Percentage of Participants | 0.0 | 0.0

6. Primary Outcome: Percentage of Participants Who Had Study Drug Discontinued Due to an AE - Double Blind Treatment Period
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. The percentage of participants who had study drug stopped during the 8-week double-blind treatment period due to an AE regardless of whether or not they completed the study was summarized by treatment arm.
Time Frame: up to Week 8
Population: All randomized participants who received at least 1 dose of study drug during double-blind treatment period.
Measure: Number; unit: Percentage of Participants
Arm/Group | L50/H12.5/A5 | L50/H12.5
Number analyzed (Participants) | 141 | 145
Percentage of Participants | 0.7 | 1.4

7. Primary Outcome: Percentage of Participants Who Experience 1 or More Adverse Events (AEs)- Long Term
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. The percentage of participants that experienced at least 1 AE during long-term period was summarized.
Time Frame: Week 9 up to Week 52 for L50/H12.5→L50/H12.5/A5 arm; Week 1 to Week 52 for L50/H12.5/A5→L50/H12.5/A5
Population: All randomized participants who received at least 1 dose of study drug during long-term reporting period.
Measure: Number; unit: Percentage of Participants
Arm/Group | L50/H12.5/A5→L50/H12.5/A5 | L50/H12.5→L50/H12.5/A5
Number analyzed (Participants) | 141 | 133
Percentage of Participants | 70.9 | 66.2

8. Primary Outcome: Percentage of Participants Who Experience 1 or More Drug-related AEs- Long Term
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. Percentage of participants that experienced at least 1 AE that was reported as possibly, probably, or definitely related to the study drug by the investigator during the long-term reporting period was summarized.
Time Frame: Week 9 up to Week 52 for L50/H12.5→L50/H12.5/A5 arm; Week 1 to Week 52 for L50/H12.5/A5→L50/H12.5/A5
Population: All randomized participants who received at least 1 dose of study drug during long-term reporting period.
Measure: Number; unit: Percentage of Participants
Arm/Group | L50/H12.5/A5→L50/H12.5/A5 | L50/H12.5→L50/H12.5/A5
Number analyzed (Participants) | 141 | 133
Percentage of Participants | 27.7 | 14.3

9. Primary Outcome: Percentage of Participants Who Experience 1 or More SAEs- Long Term
Description: An SAE is any AE occurring at any dose or during any use of Sponsor's product that does the following: results in death; is life threatening; results in persistent or significant disability/incapacity; results in or prolongs an existing inpatient hospitalization; is a congenital anomaly/birth defect; is a cancer; is associated with an overdose; is another important medical event. Those SAEs assessed as possibly, probably, or definitely related to the study drug during the long-term period were summarized.
Time Frame: Week 9 up to Week 52 for L50/H12.5→L50/H12.5/A5 arm; Week 1 to Week 52 for L50/H12.5/A5→L50/H12.5/A5
Population: All randomized participants who received at least 1 dose of study drug during long-term reporting period.
Measure: Number; unit: Percentage of Participants
Arm/Group | L50/H12.5/A5→L50/H12.5/A5 | L50/H12.5→L50/H12.5/A5
Number analyzed (Participants) | 141 | 133
Percentage of Participants | 2.1 | 3.0

10. Primary Outcome: Percentage of Participants Who Experience 1 or More Drug-related SAEs- Long Term
Description: An SAE is any AE occurring at any dose or during any use of Sponsor's product that does the following: results in death; is life threatening; results in persistent or significant disability/incapacity; results in or prolongs an existing inpatient hospitalization; is a congenital anomaly/birth defect; is a cancer; is associated with an overdose; is another important medical event. the percentage of participants that experienced an SAE that assessed as possibly, probably, or definitely related to the study drug by the investigator was summarized.
Time Frame: Week 9 up to Week 52 for L50/H12.5→L50/H12.5/A5 arm; Week 1 to Week 52 for L50/H12.5/A5→L50/H12.5/A5
Population: All randomized participants who received at least 1 dose of study drug during long-term reporting period.
Measure: Number; unit: Percentage of Participants
Arm/Group | L50/H12.5/A5→L50/H12.5/A5 | L50/H12.5→L50/H12.5/A5
Number analyzed (Participants) | 141 | 133
Percentage of Participants | 0.0 | 0.8

11. Primary Outcome: Percentage of Participants Who Had Study Drug Discontinued From the Study Due to an AE- Long Term
Description: An AE was defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the product, whether or not considered related to the use of the product. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition which was temporally associated with the use of the product, was also an AE. The percentage of participants who had study drug discontinued during the 44 week extension due to an AE regardless of completion status were summarized.
Time Frame: Week 9 up to Week 52 for L50/H12.5→L50/H12.5/A5 arm; Week 1 to Week 52 for L50/H12.5/A5→L50/H12.5/A5
Population: All randomized participants who received at least 1 dose of study drug during extension period.
Measure: Number; unit: Percentage of Participants
Arm/Group | L50/H12.5/A5→L50/H12.5/A5 | L50/H12.5→L50/H12.5/A5
Number analyzed (Participants) | 141 | 133
Percentage of Participants | 2.1 | 2.3

12. Secondary Outcome: Change in Trough Sitting Systolic Blood Pressure (SiSBP)-Double-Blind Treatment Period
Description: Sitting systolic blood pressure was measured by automated sphygmomanometer pre-dose on Day 1 (baseline) and at 24 ± 2 hours after the last study drug administration at Week 8.
Time Frame: Baseline and Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | L50/H12.5/A5 | L50/H12.5
Number analyzed (Participants) | 141 | 144
mmHg | -17.7 [-19.6 to -15.9] | -7.5 [-9.3 to -5.7]
Statistical Analysis 1: Comparison: L50/H12.5/A5 vs L50/H12.5; Test type: Superiority or Other; p < 0.001, Constrained Longitudinal Data Analysis — Model including treatment, time and the interaction of time by treatment with a restriction of the same baseline mean across treatment groups; Difference in Least Squares Means = -10.3, 95% CI 2-sided [-12.8 to -7.7]

ADVERSE EVENTS:
Time Frame: Double blind treatment period - Week 1 up to Week 8; Extension - Week 9 up to Week 52
Description: All randomized participants who received at least 1 dose of study drug during the reporting period.
Groups:
- L50/H12.5- Double Blind Treatment Period: Participants received L50/H12.5 combination tablet, orally once daily for 8 weeks
- L50/H12.5/A5 - Double Blind Treatment Period: Participants received L50/H12.5/A5 combination tablet, orally once daily for 8 weeks
- L50/H12.5/A5→L50/H12.5/A5 - Extension: Participants who received L50/H12.5/A5 combination tablet in double-blind treatment period and continued to receive L50/H12.5/A5 orally once daily for 44 weeks in extension period.
- L50/H12.5→L50/H12.5/A5 - Extension: Participants who received L50/H12.5 combination tablet in double-blind treatment period and then received L50/H12.5/A5 orally once daily for 44 weeks in extension period.
Arm/Group | L50/H12.5- Double Blind Treatment Period | L50/H12.5/A5 - Double Blind Treatment Period | L50/H12.5/A5→L50/H12.5/A5 - Extension | L50/H12.5→L50/H12.5/A5 - Extension
Serious Adverse Events (participants affected / at risk) | 2/145 | 1/141 | 2/134 | 4/133
Other Adverse Events (participants affected / at risk) | 18/145 | 10/141 | 39/134 | 42/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L50/H12.5- Double Blind Treatment Period (N=145) | L50/H12.5/A5 - Double Blind Treatment Period (N=141) | L50/H12.5/A5→L50/H12.5/A5 - Extension (N=134) | L50/H12.5→L50/H12.5/A5 - Extension (N=133)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocele (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Carcinoid tumour of the duodenum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant neoplasm of renal pelvis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L50/H12.5- Double Blind Treatment Period (N=145) | L50/H12.5/A5 - Double Blind Treatment Period (N=141) | L50/H12.5/A5→L50/H12.5/A5 - Extension (N=134) | L50/H12.5→L50/H12.5/A5 - Extension (N=133)
Nasopharyngitis (Infections and infestations) | 9 (9) | 3 (3) | 30 (35) | 30 (44)
Blood uric acid increased (Investigations) | 10 (10) | 7 (7) | 4 (5) | 7 (7)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (3) | 7 (7) | 7 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 4 (4) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication timelines.